CLINICAL TRIAL: NCT04207021
Title: Evaluation of the Effectiveness of Curcumin-based Food Supplement in Reducing Pain and Inflammatory Component in People With Osteoarthritis
Brief Title: Effectiveness of Curcumin-based Food Supplement in Reducing Pain and Inflammatory Component in Osteoarthritis
Acronym: FENOXI-1900
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KOS Care SRL - Istituto di Riabilitazione Santo Stefano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FENOXI-19
Record Dates: First submitted 2019-12-13; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Osteoarthritis; Knee Pain Chronic
Keywords: Curcumin
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): the study involves the intake of two capsules per day, one capsule to be taken before breakfast and one before dinner for a period of 6 weeks of a nutritional supplement
  INTERVENTION CAPSULE COMPOSITION active substances for 2 capsules Bio Curcumin 400 mg Polydatin 00 mg Beta-Caryophyllene 48 mg
  Interventions: Dietary Supplement: Experimental: Curcumin derivate
- placebo (Placebo Comparator): particpants included in the placebo group will take two capsules per day (containing no bioactive compound, only hydroxypropyl methylcellulose, gellan gum, pigment), one capsule to be taken before breakfast and one before dinner for a period of 6 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Experimental: Curcumin derivate — two capsules per day, one capsule to be taken before breakfast and one before dinner for a period of 6 weeks.
  Arms: intervention
Dietary Supplement: Placebo — two capsules per day (containing no bioactive compound, only hydroxypropyl methylcellulose, gellan gum, pigment), one capsule to be taken before breakfast and one before dinner for a period of 6 weeks.
  Arms: placebo

SUMMARY:
INTRODUCTION The treatment of OA is mostly symptomatic and includes the use of analgesics, NSAIDs, exercise and even surgery. However, the use of long-term NSAIDs is associated with potentially serious side effects. As a result, the use of alternative and complementary therapies (CAM), such as nutritional therapies in patients with OA, is extremely frequent.

The objective of this study will be to evaluate the effectiveness of a dietary supplement based on curcumin, polydatin and beta-caryophyllene, on the reduction of pain and inflammatory component in individuals with knee OA.

MATERIAL AND METHOD Study design Intervention study with two parallel arms, randomized, double-blind, placebo-controlled.

Study population Participants in the study will be recruited at the Santo Stefano Rehabilitation Institute. The first group will be treated with curcumin-based supplement for 6 weeks; the second group will be treated with placebo for 6 weeks.

Inclusion/exclusion criteria Inclusion criteria

* Presence of osteoarthritis of the knee. Traditional American College of Rheumatology criteria, which are based on the presence of pain (knee pain) plus at least three of the following characteristics, will be used for the diagnosis of osteoarthritis of the knee:
* Age > 50 years
* Stiffness in the morning < 30 minutes
* Presence of articular rusting
* Painfulness of the bones
* Tumefaction of the bones
* Absence of palpable heat Knee pain in this study is defined as having experienced at least moderate pain in the most affected knee (a score of 30 mm or more on an analog visual scale - VAS - as assessed by the patient) for at least 25 of the previous 30 days.

Exclusion criteria

* pregnancy and breastfeeding
* other specific contraindications/intolerances to the compound
* intake of other supplements
* treatment with anti-inflammatory or pain-relieving drugs for other clinical conditions at the time of enrolment
* Participation in other clinical studies All participants will be allowed to use analgesics (e.g. paracetamol) to control pain when needed. The patient will, however, be required to avoid / suspend the use of analgesics at least 12 hours before the baseline visit and subsequent checkups.

DETAILED DESCRIPTION:
INTRODUCTION Gonarthrosis is the most common disorder of the musculoskeletal system, with an age-related prevalence varying between 12-55%. The treatment of OA is mostly symptomatic and includes the use of analgesics, NSAIDs, exercise and even surgery. However, the use of long-term NSAIDs is associated with potentially serious side effects, with a high risk of hospitalization and death. As a result, the use of alternative and complementary therapies (CAM), such as nutritional therapies in patients with OA, is extremely frequent.

The objective of this study will be to evaluate the effectiveness of a dietary supplement based on curcumin, polydatin and beta-caryophyllene (FENOXIDOL™-Mivell), on the reduction of pain and inflammatory component in individuals with knee OA.

MATERIAL AND METHOD Study design Intervention study with two parallel arms, randomized, double-blind, placebo-controlled to assess the effectiveness of the dietary supplement in reducing perceived pain, will also be evaluated secondarily the improvement of joint function, changes in serum levels of PCR, inflammatory cytokines (TNF-alpha and IL-6) and nitrates / nitrites at the level of saliva and any change in the use of painkillers when needed.

Intervention Intervention group: the study involves the intake of two capsules per day, one capsule to be taken before breakfast and one before dinner for a period of 6 weeks.

The FENOXIDOL™ supplement and its placebo (visually identical capsules, but without active ingredients) will be supplied by the company Mivell Srls participating in the PrIntAge project. For the composition of the placebo, see the declaration attached to this document by Mivell Srls.

FENOXIDOL™ is a natural anti-inflammatory supplement designed to counteract, without any known side effects, acute and chronic inflammatory phenomena, especially those associated with joints, muscles and bones. The product has been formulated using naturally derived extracts in the quantities shown in the table below.

PHENOXIDOL CAPSULE COMPOSITION active substances for 1 capsule for 2 capsules Bio Curcumin 200 mg 400 mg Polydatin 50 mg 100 mg Beta-Caryophyllene 24 mg 48 mg

It should be noted that the product FENOXIDOL™ and its components have not been associated to date with any side effects, the active ingredients of the formula are all listed in Annex 1 of the Italian Ministry Decree of 10 August 2018 governing the use in food supplements of herbal substances and preparations as updated by Decree 9 January 2019.

It should also be noted that the FENOXIDOL™ product has no Gluten Free certification.

Placebo group: the study involves taking two capsules per day of placebo, one capsule before breakfast and one before dinner for a period of 6 weeks.

The placebo will consist of capsules with no active ingredients containing cellulose, fatty acid magnesium salts, and silicon dioxide.

All participants will be allowed to use anti-inflammatory drugs (ibuprofen up to 400 mg per 2/day) to control pain, if needed. The patient will, however, be required to avoid / suspend the use of anti-inflammatory at least 12 hours before the visit to baseline and subsequent checkups and to record the use.

Treatment, randomisation and blinding kits Mivell Srls will prepare patient kits containing treatment capsules in proportion to the time of administration and sample size considered and will send them by courier to the Pharmacy of the Istituto di Riabilitazione Santo Stefano. In order to carry out the double-blind study, these kits will be assigned, by Mivell Srls, identification codes based on the randomization lists generated by a statistical software. Blinding will be maintained for the entire duration of the study, until the analysis of the data and, possibly, interrupted only at the time of highlighting potential adverse winds in the participants.

The patient's compliance with the treatment will be calculated on the basis of the percentage of residual doses at the end of the study and on the basis of the compilation of a diary.

Biological samples and data collection Data will be collected on age, gender, educational level, BMI, employment, physical activity at work and in leisure time (IPAQ Questionnaire), tobacco habits, presence of comorbidity, type of diet (food frequency questionnaire related to the last week, with particular regard to the intake of substances with anti-inflammatory / antioxidant power, eg: seeds and dried fruit, dark chocolate, bananas, avocado, soya products, leafy vegetables, fish, garlic, curry, rosemary, ginger, saffron, (see Cavicchia, 2009), use of drugs (with particular regard to the frequency of taking painkillers and anti-inflammatory drugs in the previous six weeks) and supplements. The following will also be evaluated: duration of the disease, presence of osteoporosis, orthopaedic-neurological comorbidity, trauma, type of work, obligatory postures, use of special shoes/touches.

The objective examination will allow the evaluation of the degree of joint impairment, the completion of the WOMAC questionnaire, the pVAS scale (Visual Analogue Scale for pain), knee height from the ground, A diary of the frequency of use of pain control drugs (ibuprofen up to 400mg 2/day), to be completed by the patient or care-giver, will also be delivered.

The volume of blood collected will be 5 ml, as part of the blood sample performed for chemical and clinical tests provided for in normal clinical practice.

Blood sample testing will be performed immediately after collection at GSS Laboratories, using standard methods.

The concentration of nitrites and nitrates, IL-1 beta, IL-6 and TNF-alpha will be evaluated at the salivary level. Salivary collection will be done by means of Salivets. Dosages of nitrite and nitrate, IL-6 and TNF-alpha will be conducted on morning saliva sample. Salivary samples will be processed at the Laboratory of Molecular Biology of the Hygiene Section of the Department of Biomedical Sciences and Public Health - Polytechnic University of Marche, with delivery within the day or refrigerated for a maximum of 4 days before transport from GSS premises to the analysis laboratory.

Adverse reactions There are currently no adverse reactions associated with taking FENOXIDOL™ as a dietary supplement. However, in this study, all adverse reactions reported spontaneously by the patient or detected by the investigator will be reported on the Case Report Form (CRF).

ETHICAL AND LEGAL ASPECTS The procedures in the study regarding conduct, conduct and documentation have been prepared to ensure compliance with the ethical principles set out in the Helsinki Declaration and its revisions. The design of the research also included guidelines for Good Clinical Practice (GCP).

The study will be conducted taking into account regulatory requirements and legal requirements and the study will be initiated following the obtaining of the evaluation and approval of the study by the Regional Ethics Committee and the completion of administrative requirements provided by the institution where the study is conducted.

In addition

* Before enrolment, all potentially eligible patients should receive full information about the study;
* In order to be enrolled, patients must give their consent to the processing of personal data in anonymous and aggregate form, in accordance with the GDPR, European Regulation 679/2016 on the Protection of Personal Data.
* the patient must be informed that his or her data may be examined by authorised personnel or members of the competent ethics committee and by officials of the competent regulatory authorities
* Patient information and consent forms are included in the documentation attached to the request for approval by the Regional Ethics Committee.

References

Altman R, Alarcón G, Appelrouth D, Bloch D, Borenstein D, Brandt K, Brown C, Cooke TD, Daniel W, Feldman D, et al. The American College of Rheumatology criteria for the classification and reporting of osteoarthritis of the hip. Arthritis Rheum. 1991;34:505-14.

Arellano FM. The withdrawal of rofecoxib. Pharmacoepidemiology and Drug Safety. 2005;14(3):213-217.

Bannuru RR, Osani MC, Al-Eid F, Wang C. E Efficacy of curcumin and Boswellia for knee osteoarthritis: Systematic review and meta-analysis. Semin Arthritis Rheum. 2018 Dec;48(3):416-429.

Cavicchia PP, Steck SE, Hurley TG, Hussey JR, Ma Y, Ockene IS, Hébert JR. A New Dietary Inflammatory Index Predicts Interval Changes in Serum High-Sensitivity C-Reactive Protein1-3. The Journal of Nutrition. 2009; 139(12): 2365-72.

de Koning EJ, Timmermans EJ, van Schoor NM, Stubbs B, van den Kommer TN, Dennison EM, Limongi F, Castell MV, Edwards MH, Queipo R, Cooper C, Siviero P, van der Pas S, Pedersen NL, Sánchez-Martínez M, Deeg DJH, Denkinger MD; EPOSA Group. Within-Person Pain Variability and Mental Health in Older Adults With Osteoarthritis: An Analysis Across 6 European Cohorts. J Pain. 2018 Jun;19(6):690-698.

Felson DT, Lawrence RC, Hochberg MC, et al. Osteoarthritis: new insights-part 2: treatment approaches. Annals of Internal Medicine. 2000;133(9):726-737.

Herman CJ, Allen P, Hunt WC, Prasad A, Brady TJ. Use of complementary therapies among primary care clinic patients with arthritis. Preventing Chronic Disease. 2004;1:1-15.

Herold G. Innere Medizin. Köln: Gerd Verlag; 2007: 614-615 Jordan KM, Arden NK, Doherty M, et al. EULAR recommendations 2003: an evidence based approach to the management of knee osteoarthritis: report of a Task Force of the Standing Committee for International Clinical Studies including Therapeutic Trials (ESCISIT) Annals of the Rheumatic Diseases. 2003;62:1145-1155.

Liu X, Machado GC, Eyles JP, Ravi V, Hunter DJ. Dietary supplements for treating osteoarthritis: a systematic review and meta-analysis. Br J Sports Med. 2018 Feb;52(3):167-175.

Mobasheri A, Henrotin Y. Comment on: Efficacy of Curcumin and Boswellia for knee osteoarthritis: Systematic review and meta-analysis. Semin Arthritis Rheum. 2018 Apr 11.

Moskowitz RW, Abramson SB, Berenbaum F. Coxibs and NSAIDs-clearing the air. Osteoarthritis and Cartilage. 2005;13(7):545-547. [PubMed] National Institute of Arthritis and Musculosceletal and Skin Diseases. Handout on Health: Osteoarthritis. May 2016. Available at http://www.niamsnihgov/Health_Info/Osteoarthritis/defaultasp.

Oliviero F, Scanu A, Zamudio-Cuevas Y, Punzi L, Spinella P. Anti-inflammatory effects of polyphenols in arthritis. J Sci Food Agric. 2018 Mar;98(5):1653-1659.

Sangha O. Epidemiology of rheumatic diseases. Rheumatology. 2000;39(supplement 2):3-12. [PubMed] World Health Organization Department of Reproductive Health and Research (WHO/RHR) and Johns Hopkins Bloomberg School of Public Health/Center for Communication Programs (CCP), Knowledge for Health Project. Family Planning: A Global Handbook for Providers (2018 update). Baltimore and Geneva: CCP and WHO, 2018.

Zhang G, Cao J, Yang E, Liang B, Ding J, Liang J, Xu J. Curcumin improves age-related and surgically induced osteoarthritis by promoting autophagy in mice. Biosci Rep. 2018 Jul 2;38(4).

Zhao P, Cheng J, Geng J, Yang M, Zhang Y, Zhang Q, Wang Y, Lu B. Curcumin protects rabbit articular chondrocytes against sodium nitroprusside-induced apoptosis in vitro. Eur J Pharmacol. 2018 Jun 5;828:146-153.

ELIGIBILITY:
Inclusion Criteria:

* Presence of osteoarthritis of the knee. Traditional American College of Rheumatology criteria, which are based on the presence of pain (gonalgia) plus at least three of the following characteristics, will be used for the diagnosis of osteoarthritis of the knee:
* Age > 50 years
* Stiffness in the morning < 30 minutes
* Presence of articular rusting
* Painfulness of the bones
* Tumefaction of the bones
* Absence of palpable heat

Exclusion Criteria:

* - pregnancy and breastfeeding (if the potential participant does not declare to be in a menopausal state)
* other specific contraindications/intolerances to the compounds contained in the supplement (e.g. celiac disease, allergy)
* simultaneous intake of other supplements
* to be at the time of enrolment for treatment with anti-inflammatory or pain-relieving treatment for other clinical conditions
* Participation in other clinical studies
* State of inability to understand or desire

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2019-12-18 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
- variation in the level of joint function measured by the Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 0, 6 weeks
  WOMAC scale is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties
  The test questions are scored on a 0-4 scale, corresponding to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up; higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations

SECONDARY OUTCOMES:
- variation of serum levels of C-reactive Protein (CRP) | 6 weeks
  Serum CRP levels were assessed by means of a commercially available CRP enzyme immunoassay
- variations of saliva levels of TNF-alpha, IL-1beta, IL-6, nitrates/nitrites | 6 weeks
  Levels of TNF-alpha, IL-1beta, IL-6, nitrates/nitrites will be evaluated by means of ELISA-testing
- variation in the use of painkillers | 6 weeks
  Painkillers utilization will be registered on a daily basis by participants, indicating dosage and daily frequency of use.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Frascarello, MD, Principal Investigator — Istituto Santo Stefano